CLINICAL TRIAL: NCT07108322
Title: Clinical Evaluation of Digital Versus Conventional Impression in Edentulous Patients With Flabby Ridge. A Randomized Controlled Clinical Trial
Brief Title: Digital Versus Conventional Impression in Edentulous Patients With Flabby Ridge.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Delta University for Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: FODMRC-2023-00111
Record Dates: First submitted 2025-08-04; First posted 2025-08-07 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-07

CONDITIONS: Flabby Ridge; Edentulous Alveolar Ridge
Keywords: Flabby ridge; Edentulous; Maxillary; digital scanning
MeSH Terms: conditions — Mouth, Edentulous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Edentulous maxillary arch with flabby ridge (Other): Conventional impression followed by intraoral scanning
  Interventions: Other: Intraoral scanning

INTERVENTIONS:
Other: Intraoral scanning — Adigital impression with intraoral scanning

SUMMARY:
The main goal of complete denture prosthodontics is to restore function, comfort, and aesthetics by replacing missing teeth and supporting structures. Flabby ridges, defined as mobile soft tissue on the alveolar ridge, pose challenges in creating stable dentures, as these tissues can displace under occlusal forces, compromising retention and support. Special impression techniques are necessary to manage flabby ridges effectively One widely accepted method is the window technique, which uses double spacers and window in the flabby tissue area. However, this technique is technically complex. This RCT aims to evaluate whether intraoral scanning (IOS) provides an alternative to the window technique for recording maxillary flabby ridges.

The hypothesis was that IOS will demonstrate superior clinical results in terms of both Retention and Patient satisfaction compared to the conventional window technique impression (WTI).

DETAILED DESCRIPTION:
Participants and setting A total of 26 participants who met all pre-defined inclusion criteria were consecutively enrolled in the study. All eligible patients presenting to the outpatient clinic at the Department of Prosthodontics, Delta University for Science and Technology, during the defined recruitment period were screened for inclusion.

Design The study utilized a crossover design, where participants were randomly assigned to receive complete dentures fabricated by using two different techniques for complete denture fabrication: Group I dentures were fabricated using the conventional window technique impression and Group II denture were fabricated using Digital impression technique. A new complete denture was delivered for each participant after 6 months, with those initially receiving Group I dentures transitioning to Group II dentures, and vice versa.

Randomization The randomization sequence was generated by a statistician using a computer-generated list of random numbers at a 1:1 allocation ratio, independent of the study's clinical team. A non-clinical assistant, who was not involved in patient recruitment or assessment, prepared the opaque, sequentially numbered, sealed envelopes and was responsible for their safekeeping in a locked cabinet. The Principal Investigator (D.E.) was responsible for screening and enrolling eligible participants. Assignment was performed by an independent dental assistant immediately prior to implementing the assigned impression technique by opening the next sequential envelope, thus ensuring adequate allocation concealment.

Interventions For Group I dentures, Window Technique Impression was employed to make the final impression, and the sequence of steps was as follows: The primary alginate impression of the edentulous maxilla was made with stock edentulous trays. Anterior maxillary flabby tissue was palpated and identified intraorally using large ball burnisher and outlined with an indelible pencil. The impression was repositioned in the patient's mouth and the markings made with an indelible pencil were transferred onto the impression surface. The impression was then poured using Type III dental stone, and one sheet of modeling wax was adapted as a spacer.

Border molding of the custom trays were made using tracing compound to capture functional extension. Then the custom tray was opened in the area of flabby tissues guided by the indelible pencil marks on the primary cast. Zinc oxide eugenol paste was loaded onto the tray to record the non-flabby tissues, ensuring detailed and stable impressions of these areas. A light coat of impression plaster was applied on the flabby ridge area using a small brush through the window area. Because the window exposes the flabby tissue, plaster captures its detail without compressing or displacing it, thereby preventing dislodgement of the denture during function and improving stability. The window technique impression was then scanned using a desktop extra-oral scanner. The scanner is equipped with four 5 MP cameras and Blue LED Multi-line technology, achieving an accuracy of 5 μm (ISO) / 8 μm. Prior to analysis, artifacts such as air bubbles and voids on the palatal surface of the WTI models were digitally removed to fabricate a 3D-printed model.

For Group II dentures, a digital impression of maxillary arch was made using an IOS to obtain the test files. Specialized soft tissue scan retractor was constructed with a resilient yet sufficiently rigid framework to fit into the vestibular area, allowing unobstructed movement of the scan head which is essential for obtaining precise intraoral data without soft tissue interference.16 Before scanning, a meticulous cleansing of the edentulous ridge was performed, followed by the removal of any residual saliva.

The scanning process for the maxillary arch started at the ridge's crest on one side and proceeded along the residual ridge until reaching the canine-incisor region. At this point, a zig-zag scanning pattern was performed to capture both the crest and the anterior palatal slope. The pathway then continued in a straight line along the ridge's crest to the other side. Subsequently, the scanner head was turned to capture the buccal aspect, moving in a straight line to the opposite buccal side. Scanning then covered the palatal incline of the tuberosity and advanced anteriorly along the posterior palatal incline until it reached the previously scanned anterior palatal slope. Finally, scanning continued in a backward direction across to the opposite side, ensuring complete coverage of the entire palatal region. The systematic scanning pathway used for all cases is important for the creation of accurate digital models that form the basis of manufactured prosthesis.

Diagram for the scanning pathway employed The resultant STL files of the scan of the window technique impression and the IOS of the maxillary arch were exported to a RapidShape D30 2016 3D-printer to produce 3D-printed models of the maxillary arch. The 3D-printed models were then duplicated by enclosing the models within a mold box ensuring it is positioned securely. Silicone molding material was mixed and poured into the box completely encasing the 3D-models until the silicone was cured. The 3D-printed cast was carefully removed from the silicone mold. Type III dental stone was mixed and poured into the silicone mold ensuring it filled all fine details and allowed to harden completely.

3D-printed cast duplicated into stone cast For both Groups, the final impression of the mandibular arch was made using border molding with green stick compound and Zn oxide and eugenol final impression material. All the conventional steps of complete denture construction then proceeded. . After the initial wax-up, the denture was verified in the patient's mouth before being processed using the compression molding technique with conventional heat-cured acrylic resin. The dentures for both groups (Conventional and Digital) were fabricated by a single, experienced dental technician. The technician was not blinded to the impression type but was instructed to use identical materials and processing techniques for the final dentures. The IOS operator (D.E.) had extensive prior experience before the trial commenced, thereby minimizing the impact of the learning curve on the results. A single operator performed all scans to reduce inter-operator variability.

On the day of denture delivery, the complete denture was checked for fit, borders, extensions and occlusion. Group I dentures were delivered to the patients. After 6 months of functional denture use and a washout period of 48 hours, Group II dentures were delivered.

Outcomes The primary endpoint of this crossover trial is the difference between the two techniques (Digital vs. Conventional) in OHRQoL as measured by the OHIP-EDENT-19 questionnaire at T0, T3 and T6. The secondary endpoint is the difference in maxillary denture retention at the same time points.

Each patient was asked to fill a questionnaire at T0 and T3, T6. OHIP-EDENT-19 was used to assess the OHRQoL. We used the Arabic version of OHIP-EDENT-19, whose psychometric properties in completely edentulous older adults have been validated. The profile consisted of 19 questions, each with a score of 0 to 4 (impaired) on the Likert scale The denture retention was measured at T0, T3, and T6 by a digital force gauge device, which measures tension or compression force (pull/push) to values up to 980 N. The snap loop of the device engaged a screw that was fixed to the geometric center of the denture bases with self-curing acrylic resin to avoid heat-induced distortion of the denture base, thus maintaining the integrity of the base adaptation. The geometric center is typically located by marking the midline of the maxillary cast, drawn from the center of the incisive papilla extending posteriorly to the midpoint of a line connecting the two hamular notches. The midpoint on this midline represents the geometric center of the maxillary arch. This point is used as a stable and balanced reference for placing attachments or screws.

The rigor of the outcome measurement for denture retention was ensured by following a standardized, quantifiable methodology utilizing a digital force gauge. Retention was evaluated by performing five consecutive pulls at each designated time point. For each pull, the peak dislodging force (the maximum resistance recorded before complete displacement) was registered by the gauge. A rest interval of 60 seconds was enforced between each pull, allowing for soft tissue recovery and the re-establishment of the crucial salivary film required for reliable physical retention measurement. The retention force was applied to a custom-fabricated attachment loop on the denture and pulled by the force gauge in a vertical direction, directly opposite to the denture's path of insertion. To eliminate kinetic or inertial errors, the force was applied at a constant, slow rate of approximately 50 mm/minute until dislodgement. Finally, the reported retention value for each time point was calculated as the mean (average) of the peak forces recorded from the five consecutive pulls, which is a common practice to minimize measurement variability and ensure the final reading is highly representative of the prosthetic retention. The device was used within its manufacturer-recommended calibration cycle to ensure accurate measurement. The instrument was newly calibrated prior to the start of the trial.

A single, calibrated examiner performed all measurements; thus eliminating inter-examiner variability. The intra-examiner reliability was assessed prior to the study using the Intra-class Correlation Coefficient (ICC), which showed high reliability (ICC > 0.90).

Statistics A statistical analysis plan was performed. Comparison between groups was made using paired t-test, while comparison between different time points was performed by using Repeated Measures ANOVA test followed by Tukey's Post Hoc test. The significant level was set to be at P ≤ 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Completely edentulous patients with maxillary flabby ridge
* Absence of infectious diseases
* Systemic good health (ASA-1/ASA-2)
* Age between 50 and 75 years
* Willingness to cooperate throughout the data collection process.

Exclusion Criteria:

* Presence of any remaining teeth
* Inability to comprehend the study's objectives and procedures
* ridge defect or lesion
* Postoperative scarring on the ridge
* Limitations in mouth opening.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2023-03-30 (Actual); Primary Completion 2025-04-29 (Actual); Study Completion 2025-06-25 (Actual)

PRIMARY OUTCOMES:
patient satisfaction | Baseline, 3 months and 6 months
  A questionnaire will be provided to score Oral Health Related Quality of Life . The scoring system used a Likert scale where a lower score indicates a better perceived quality of life, as the minimum possible score is 0 and the maximum is 76 (higher score indicating more impairment).

SECONDARY OUTCOMES:
Retention | Baseline, 3 months and 6 months
  The denture retention was measured by a digital force gauge device, which measures tension or compression force (pull/push) to values up to 980 N.

CONTACTS AND LOCATIONS:
Overall Officials: Dina M. ElAwady, PHD, Principal Investigator — Associate Professor of Prosthodontics
Locations (1):
- Delta University for Science and Technology, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No
Till the article is published